CLINICAL TRIAL: NCT05484648
Title: Dexamethasone or Dexmedetomidine as Adjunct in Fascia Iliaca Block During Positioning for Sub-arachnoid Block & Post-operative Analgesia After Femur Neck Fracture Surgery: A Randomized Control Trial
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Aga Khan University Hospital, Pakistan (Other)
Responsible Party: Principal Investigator, Haris Sheikh, Post-Graduate Trainee, Department of Anaesthesiology, Aga Khan University Hospital, Pakistan
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 7886
Record Dates: First submitted 2022-07-24; First posted 2022-08-02 (Actual); Last update posted 2022-08-02 (Actual); Status verified 2022-07

CONDITIONS: Post Operative Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Dexamethasone; Dexmedetomidine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group A (Experimental): Patients allocated to group A will receive ultrasound guided FICB with 0.375% ropivacaine 38 cc along with 8 mg dexamethasone in 2cc making a total injection volume of 40 cc.
  Interventions: Drug: Dexamethasone
- Group B (Experimental): Patients allocated to group B will receive ultrasound guided FICB with 0.375% ropivacaine 38 cc along with 1 µg/kg dexmedetomidine in 2cc dilution making a total injection volume of 40 cc.
  Interventions: Drug: Dexmedetomidine
- Group C (No Intervention): Patients allocated to group C will receive ultrasound guided FICB with 0.375% ropivacaine 38 cc along with 2 cc normal saline making a total injection volume of 40 cc. This will serve as the control arm.

INTERVENTIONS:
Drug: Dexamethasone — Dexamethasone has been used to generally favorable results in peripheral nerve blocks as adjunct. Several studies have reported prolongation in the duration of ropivacaine, mepivacaine and bupivacaine when used in combination with dexamethasone.
  Various mechanisms for the beneficial adjunctive effect of dexamethasone with Local Anesthetics (LA) have been proposed. One theory suggests that the improved analgesia and increased blockade duration is due to its anti-inflammatory properties. It also acts as a local vasoconstrictor and thus may act by reducing LA absorption. Furthermore, it also increases the activity of inhibitory potassium channels on nociceptive C-Fibers.
  Arms: Group A
Drug: Dexmedetomidine — Dexmedetomidine is another promising drug being used as a local anaesthetic adjuvant in peripheral nerve blocks. It is an alpha-2 agonist, which has shown to have prolonged duration of postoperative analgesia when given with LA for peripheral nerve blocks with other beneficial effects such as reducing the opioid consumption. Alpha-2-agonists such as dexmedetomidine cause hyperpolarization-activated cation currents which inhibit the transmission of nociceptive fibers.
  Arms: Group B

SUMMARY:
Femur fracture is a common injury occurring in the young due to trauma as well as amongst the elderly due to fall. Reduction and fixation of femur fractures pose a challenge to the anesthesiologist. These fractures are intensely painful as the pain arises from the periosteum and even slight movement can cause muscle forces to angulate and deform the fractured fragments which apart from causing extreme pain also make the reduction of the fracture quite difficult. Sub-arachnoid block (SAB) is a commonly used technique for lower-limb surgeries. It provides excellent surgical anesthesia and is a largely safe and reliable anesthetic technique. However, for femur fracture repair, positioning the patient for SAB not only causes extreme pain but it also makes administration of SAB difficult due to inappropriate position. Another limitation of SAB is its limited duration of action. Hence, conventional pain management modalities which include opioids and NSAIDs are used to manage pain before and during the administration of SAB and during the post-operative period. These conventional pain management drugs are associated with significant adverse effects and should be used with caution especially in the elderly with multiple comorbids.

Recently, fascia iliaca block (FICB) has been used not only as part of multi-modal peri-operative analgesic regime for femur fractures but also to provide adequate analgesia for appropriate SAB positioning. FICB fills the plane underneath the fascia iliaca with local anesthetic and acts on the femoral, lateral femoral cutaneous and obturator nerves and thus provides adequate analgesia for femur fractures for up to 24-48 hours. FICB is also associated with less side effects when compared to conventional pain management modalities and provides adequate unilateral analgesia with fewer autonomic and neurological complications when compared with epidural analgesia.

Traditionally, local anesthetics have been used for most of the peripheral nerve blocks (PNB), however multiple adjuncts such as opioids, ketamine and clonidine have been used to prolong the duration of action as well as decrease the local anesthetic dosage. Among the adjuncts, dexamethasone has been used to generally favorable results in PNBs. Dexmedetomidine is another promising drug being used as a local anaesthetic adjuvant in peripheral nerve blocks. It is an alpha-2 agonist, which has shown to have prolonged duration of postoperative analgesia when given with LA for peripheral nerve blocks with other beneficial effects such as reducing the opioid consumption.

In this study, the investigators compare dexamethasone with dexmedetomidine as an adjunct when combined with ropivacaine in FICB.

ELIGIBILITY:
Inclusion Criteria:

* Age group (18-80)
* Undergoing elective/emergency femur fracture repair under sub-arachnoid block
* ASA status I-III

Exclusion Criteria:

* Participation in any other trial
* Known hypersensitivity to study medications
* Seizure disorder
* Coagulation disorder
* Infection over injection site
* Hemodynamic Instability
* Concurrent medications use that is contraindicated with study medications

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-01-01 (Estimated); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Pain score after fascia iliaca block placement | Static Pain at 5 minutes after placement of block.
  Static pain will be recorded at 5 minute interval with the help of Numeric Rating Scale (NRS) of 0 to 10 (with 0 being no pain at all and 10 being worst imaginable pain).
Pain score after fascia iliaca block placement | Static Pain (at 10 minutes after placement of block.
  Static pain will be recorded at 10-minute interval with the help of Numeric Rating Scale (NRS) of 0 to 10 (with 0 being no pain at all and 10 being worst imaginable pain).
Pain score during positioning of patient for sub-arachnoid block | Dynamic Pain during positioning for sub-arachnoid block
  After 15 minutes of fascia iliaca block placement, patients will be positioned for sub-arachnoid block. At this point, dynamic pain will be recorded with the help of Numeric Rating Scale (NRS) of 0 to 10 (with 0 being no pain at all and 10 being worst imaginable pain).

SECONDARY OUTCOMES:
Duration of postoperative analgesia | Till 24 hours post surgery
  This will be measured by the demand to first rescue analgesic
Post-operative Pain | Arrival in PACU (0 hours)
  Post-operative pain will be assessed via the Numeric Rating Scale (NRS) of 0 to 10 (with 0 being no pain at all and 10 being worst imaginable pain).
Post-operative Pain | 6 hours after surgery
  Post-operative pain will be assessed Numeric Rating Scale (NRS) of 0 to 10 (with 0 being no pain at all and 10 being worst imaginable pain).
Post-operative Pain | 12 hours after surgery
  Post-operative pain will be assessed via the Numeric Rating Scale (NRS) of 0 to 10 (with 0 being no pain at all and 10 being worst imaginable pain).
Post-operative Pain | 24 hours after surgery
  Post-operative pain will be assessed via the Numeric Rating Scale (NRS) of 0 to 10 (with 0 being no pain at all and 10 being worst imaginable pain).
Patient Satisfaction | 24 hours after surgery
  Patient satisfaction would be assessed via the Likert Scale

CONTACTS AND LOCATIONS:
Overall Officials: Samie Asghar, MBBS, FCPS, Principal Investigator — Aga Khan University

IPD SHARING:
Plan to Share IPD: No